CLINICAL TRIAL: NCT01604187
Title: Procedural Pain Treatment With Transmucosal Sublingual Fentanyl Tablet in Colonoscopy Patients
Acronym: Abstral
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Turku University Hospital (Other Government)
Responsible Party: Principal Investigator, Mari Fihlman, MD, Turku University Hospital
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Supportive Care
Other Study IDs: Abstral
Record Dates: First submitted 2012-05-21; First posted 2012-05-23 (Estimated); Last update posted 2019-09-11 (Actual); Status verified 2019-09

CONDITIONS: Colonoscopy; Pain
Keywords: sublingual fentanyl; pain in coloscopy; The efficacy and safety of fentanyl transmucosal tablet to placebo in patients having colonoscopy.
MeSH Terms: conditions — Pain | interventions — Fentanyl

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fentanyl (Active Comparator): Ten minutes before the procedure fentanyl 100 mikrograms sublingual tablet will be given to the patient.
  Interventions: Drug: Fentanyl
- Placebo (Placebo Comparator): Ten minutes before the procedure placebo sublingual tablet will be given to the patient.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Fentanyl — Ten minutes before the procedure fentanyl sublingual tablet (Abstral ® 100 µg, ProStrakan) will be given to the patient.
  Arms: Fentanyl
Drug: Placebo — Ten minutes before the procedure placebo sublingual tablet will be given to the patient.
  Arms: Placebo

SUMMARY:
Colonoscopy is generally considered an invasive procedure that causes remarkable pain to the patient. The pain associated with the procedure is not caused by the insertion of the scope but from inflating of the colon in order to do the inspection. It has been shown that colonoscopy can be performed successfully without sedation (Leung, 2010), but many patients feel discomfort during the procedure. Factors predicting a painful colonoscopy are female-gender, degree of patient nervousness and the technical difficulty of the colonoscopy (Ylinen et al. 2009). Also age under 40, previous abdominal surgery and use of sedation are associated with painful colonoscopy ( Seip et al. 2009). Most often sedation and/or analgesia are achieved by administering a benzodiazepine or a combination of a benzodiazepine and an opioid (Fanti et al. 2009, Maskelar et al. 2009,), dexmedetomidine (Dere et al. 2009) or by using non-pharmacologic methods (Amer-Cuenca et al. 2011). Tramadol as monotherapy did not significantly decrease pain intensity or endoscopist's evaluation of colonoscopy (Grossi et al. 2004). Currently, intravenous midazolam is the drug used most commonly to introduce some sedation for colonoscopy. Intravenous sedation definitely increases the cost of procedure; drug administration, need for pulse oximetry monitoring and the need for follow-up after the procedure make colonoscopy sometimes expensive and troublesome. It has also been shown, that low-dose midazolam neither relieves discomfort nor makes patients forget it (Elphick et al. 2009).

Fentanyl is a short-acting opioid widely used in anesthesia management. Transmucosal sublingual formulation of fentanyl has been developed to further improve the management of pain. When administered as a sublingual fast-dissolving tablet (Abstral®) that is placed under the tongue, the effects is fast and predictable. Its active ingredient is absorbed by the body through the mucous membrane. After administration of buccal fentanyl maximum plasma drug concentration was measured after 25 minutes (Darwish et al. 2011). Plasma fentanyl concentrations versus time following buccal and sublingual administration are very similar (Darwish et al. 2008). Abstral® sublingual tablets should be administered directly under the tongue at the deepest part. Sublingual administration is an easy and non-invasive method of pain treatment for the patient coming to colonoscopy done as an office based procedure. Other advantages compared to invasive methods are improved comfort of patients and no need for intravenous access because of pain relief. Before, it has been used in the management of breakthrough pain in cancer patients. Sublingual fentanyl is shown to be effective and well-tolerated for the treatment of breakthrough cancer pain (Uberall et al. 2011). The use of transmucosal tablet for colonoscopy patients is a quite new approach.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the efficacy of fentanyl transmucosal tablet to placebo in patients having colonoscopy.

Fentanyl is a highly lipophilic drug absorbed very rapidly through the oral mucosa and more slowly through the gastrointestinal tract. Orally administered fentanyl undergoes pronounced hepatic and intestinal first pass effects.

Abstral® is a quick dissolving sublingual tablet formulation. Rapid absorption of fentanyl occurs over about 30 minutes following administration of Abstral®. The bioavailability of Abstral® has not been studied but is estimated to be about 70%. Mean maximal plasma concentrations of fentanyl range from 0.2 to 1.3 ng/ml (after administration of 100 to 800 µg Abstral®) and are reached within 22.5 to 240 minutes.

Fentanyl is metabolised primarily via CYP3A4 to a number of pharmacologically inactive metabolites, including norfentanyl. Within 72 hours of intravenous fentanyl administration around 75% of the dose is excreted into the urine, mostly as metabolites, with less than 10% as unchanged drug. About 9% of the dose is recovered in the faeces, primarily as metabolites. Total plasma clearance of fentanyl is about 0.5 l/h/kg. After Abstral® administration, the main elimination half-life of fentanyl is about 7 hours (range 3-12.5 hours) and the terminal half-life is about 20 hours (range 11.5-25 hours). Impaired hepatic or renal function could cause increased serum concentrations. Elderly, cachectic or generally impaired patients may have a lower fentanyl clearance, which could cause a longer terminal half-life for the compound.

This is a randomized controlled double-blind study. A total of 200 patients will be included. The patients are recruited from 18-85 year old male or female patients undergoing colonoscopy. In view of previous studies (Amer-Cuenca et al. 2011) it can be calculated that 87 patients will be needed per group to demonstrate a 30% decrease in the worst experienced pain at a level of significance P = 0.05 and power of 90%. Because of possible dropouts, 100 patients will be recruited to both groups. Pain will be assessed by numeral rating scale (NRS). For the calculation of the sample size, coefficient of variation is assumed to be 70% in both groups.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-III
* Colonoscopy
* Written informed consent from participating subject

Exclusion Criteria:

* A previous history of intolerance to the study drug or related compounds and additives
* History of alcoholism, drug abuse, psychiatric, psychological or other emotional problems that are likely to invalidate informed consent
* Sleep apnoea
* Chronic obstructive pulmonary disease
* BMI ≥ 35 or weight < 50 kg
* SpO2 < 90 %
* Concomitant drug therapy known to cause significant enzyme induction or inhibition of CYP 3A4.
* Pregnancy or nursing.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Actual)
Dates: Start 2012-04; Primary Completion 2019-04-22 (Actual); Study Completion 2019-04-30 (Actual)

PRIMARY OUTCOMES:
Efficacy of fentanyl transmucosal tablet to placebo in patients having colonoscopy.
  Anxiety will be measured using NRS (0 = no anxiety, 10=maximal anxiety). Pain will be monitored by using numercal rating scale NRS (0-10), sedation by using NRS (0-10, 0= not sedated at all, 10=no response) . Nurse's and surgeon's satisfaction with the procedure will be evaluated using NRS (0-10). Adverse effects of opioids will be evaluated by patients using NRS (0-10)) for the following items: drowsiness (alert / very drowsy), pleasantness (very unpleasant / very pleasant feeling) and nausea/vomiting (no nausea / very strong nausea). In addition, all other adverse effects will be recorded.

SECONDARY OUTCOMES:
The safety of fentanyl transmucosal tablet to placebo in patients having colonoscopy.
  SpO2 and breath rate will be followed throughout the procedure. If the peripheral arterial oxygen saturation decreases below 90 % or breath rate falls below 8 per min, additional oxygen will be given. In case of excess opioid effects, naloxon 0.1mg iv will will be given.
  The patients will be interviewed by telephone on the first day after the procedure approximately 24 hours later and.

CONTACTS AND LOCATIONS:
Overall Officials: Klaus T Olkkola, professor, Principal Investigator — Turku University Hospital
Locations (1):
- Turku University Hospital, Turku, Finland